CLINICAL TRIAL: NCT04248205
Title: Intra-operative Use of Ketamine for Post-Operative Analgesia in Patients Undergoing Hemorrhoidectomy: A Prospective, Randomized Controlled Trial.
Brief Title: Ketamine for Post-operative Analgesia in Hemorrhoidectomy
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11475
Record Dates: First submitted 2020-01-27; First posted 2020-01-30 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Hemorrhoids
Keywords: hemorrhoidectomy; ketamine; post operative pain
MeSH Terms: conditions — Hemorrhoids; Pain, Postoperative | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intraoperative ketamine infusion (Active Comparator): Subjects in this group will receive standard anesthesia during surgery and a dose of ketamine at 0.3 mg/kg IV bolus prior to surgical incision. If the procedure lasts more than 1 hour, an additional bolus dose will be given.
  Interventions: Drug: Ketamine
- Control group (No Intervention): This group will only receive the standard anesthesia during surgery with no ketamine.

INTERVENTIONS:
Drug: Ketamine — Standard general anesthesia PLUS ketamine will be given for post-operative analgesia
  Arms: Intraoperative ketamine infusion

SUMMARY:
This is a prospective, randomized study of ketamine versus no ketamine in approximately 100 patients undergoing hemorrhoidectomy for Grade III or IV hemorrhoids. The participants will be blinded to which treatment arm they are assigned, because participants will be under anesthesia when the ketamine is administered. The investigators will know whether the participant receives ketamine or not.

DETAILED DESCRIPTION:
Participants will be randomized into 2 groups: intraoperative ketamine infusion during operation or routine anesthesia with no ketamine. Participants are pre-medicated in the operating room with the same regimen: Gabapentin 300mg, Ultram 50mg, and Tylenol 1000mg.

For participants in the ketamine group, a pain dose of ketamine 0.3mg/kg IV bolus dosing will be given prior to incision. If the procedure lasts longer than 1 hour, an additional bolus dose will be given. All participants will undergo general anesthesia and receive routine anesthesia care, aside from ketamine verus no ketamine. All participants will also receive standard local anesthesia including a local regional perianal nerve block.

The procedure will be performed by three different surgeons, with the surgery done the same way using ligasure hemorrhoidectomy. Participants will all be sent home with the same post-operative instructions and pain medications to include: Tylenol 1000mg, oxycodone 5mg, ibuprofen 800mg, fiber/miralax, and tub baths twice daily for 15 minutes.

A patient pain handout will be given to participants upon discharge with instructions to rate pain according to a numeric rating scale and the Wong-Baker FACES pain scale. Participants will be contacted by a member of the research team to assess their post-operative pain based on a numeric rating scale. All participants will undergo post-operative clinic follow-up at 2 weeks post-operation. At that time they will be instructed to bring their oxycodone bottle to assess how many pills the participant required. The clinic medical assistant will count the number of remaining pills and record this in the electronic medical record. If a participant forgets their pain scale record or medications, a post-operative phone interview will be performed after the clinic appointment to gather this information.

The investigators will randomize 50 participants to the ketamine group and 50 participants to the placebo group. Study will take place until all participants have been analyzed, approximately 8-12 months. Randomization will occur using a statistical method with study arms placed into individual envelopes that will be stored at the University of Oklahoma (OU) Surgery Center. The investigator will blindly pull an envelope from the stack which will identify the participant's treatment arm. The participants will be blinded and not informed of their arm of the study as to not create bias toward subjective pain. Practitioners will not be blinded for ease of medication administration. The procedures will occur at OU Surgery Center by one of three surgeons. Anesthesiologists will administer ketamine based on study arm.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-100
* Undergoing a hemorrhoidectomy for Grade III or IV hemorrhoids.

Exclusion Criteria:

* Inability to undergo general anesthesia
* Contraindications to hemorrhoidectomy
* History of schizophrenia or other hallucinatory psychiatric illnesses
* History of psychosis
* Chronic narcotic usage defined as either having a pain contract with a pain management specialist and no narcotic usage for one month prior to hemorrhoidectomy.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-06-15 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Change in post-operative narcotic usage | two weeks post-operation
  Standardized pain control regimen with ketamine; at two week surgical follow-up visit patient will bring their oxycodone prescription and we will count the number of pills that were taken.

SECONDARY OUTCOMES:
Change in post-op pain | Post-op days 1, 3, 5, 7, and 10
  Wong-Baker FACES Pain Rating Scale, which ranges from 0 to 10, with 0 being represented by a happy face indicating "No Hurt" to 10, represented by a crying face, indicating "hurts like the worst pain imaginable".

CONTACTS AND LOCATIONS:
Overall Officials: Steven N Carter, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Himmelseher S, Durieux ME. Ketamine for perioperative pain management. Anesthesiology. 2005 Jan;102(1):211-20. doi: 10.1097/00000542-200501000-00030. No abstract available. PMID 15618805
- [Background] Gorlin AW, Rosenfeld DM, Ramakrishna H. Intravenous sub-anesthetic ketamine for perioperative analgesia. J Anaesthesiol Clin Pharmacol. 2016 Apr-Jun;32(2):160-7. doi: 10.4103/0970-9185.182085. PMID 27275042
- [Background] Luggya TS, Roche T, Ssemogerere L, Kintu A, Kasumba JM, Kwizera A, Tindimwebwa JV. Effect of low-dose ketamine on post-operative serum IL-6 production among elective surgical patients: a randomized clinical trial. Afr Health Sci. 2017 Jun;17(2):500-507. doi: 10.4314/ahs.v17i2.25. PMID 29062346